CLINICAL TRIAL: NCT00438100
Title: Randomized Control Study of Capecitabine vs. S-1 in Unresectable or Recurrent Breast Cancer Patients
Brief Title: Capecitabine vs. S-1 in Unresectable or Recurrent Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Japan Breast Cancer Research Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JBCRN-05; UMIN000000609 (Registry Identifier: UMIN CTR)
Record Dates: First submitted 2007-02-18; First posted 2007-02-21 (Estimated); Results first posted 2015-05-29 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Breast Neoplasms
Keywords: Breast Neoplasms; Drug Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; S 1 (combination); titanium silicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Capecitabine arm (Active Comparator): Capecitabine (Xeloda): 1600 mg/m2 orally bid daily for day 1 through day 21 followed by 7-day washout; repeat this as a course.
  Interventions: Drug: Capecitabine
- S-1 arm (Experimental): S-1: 80 mg/m2 orally bid daily for day 1 through day28 followed by 14-day washout; repeat this as a course.
  Interventions: Drug: S-1

INTERVENTIONS:
Drug: Capecitabine — 1600 mg/m2 orally bid daily for day 1 through day 21 followed by 7-day washout; repeat this as a course.
  Other Names: Xeloda
  Arms: Capecitabine arm
Drug: S-1 — 80 mg/m2 orally bid daily for day 1 through day 28 followed by 14-day washout; repeat this as a course.
  Other Names: TS-1
  Arms: S-1 arm

SUMMARY:
To investigate and compare the efficacy and safety of S-1 vs. Capecitabine as primary chemotherapy in patients with inoperable or recurrent breast cancer.

DETAILED DESCRIPTION:
The incidence of breast cancer is increasing in Japan: 33,676 women were diagnosed with breast cancer in 2001, making it the leading cause of cancer among women since 1995. Statistical database in Exel format/outline of health welfare statistics from the Ministry of Labor, Health, and Welfare show that the number of deaths from breast cancer was 9,806 in 2003. Because the ten-year survival rate is about ninety percent in Stages 0 and I breast cancer patients, detection and treatment at an earlier stage can lead to higher survival rates. However, the recurrence rate increases as the disease progresses. In addition, about thirty percent of all breast cancer patients are believed to have recurrent disease. Thus, developing treatments against recurrence may be an important task.

The Guideline for Breast Cancer Treatment, 2004 version, recommends chemotherapy, including anthracyclines or taxanes as a first-line chemotherapy for metastatic or recurrent (grade B recommendation) breast cancer. In a second-line therapy recommended for metastatic or recurrent diseases, the Guideline reports that a combination of capecitabine, a 5Fu derivative (an oral chemotherapy of pyrimidine fluorides approved in 2003) with docetaxel is superior to docetaxel alone for improving survival. This regimen is recommended for patients with cardiac malfunction who cannot be treated with anthracyclines (grade B recommendation). However, data are lacking to support capecitabine as a standard regimen as a second-line therapy; its efficacy needs verification and further study. Accordingly, this study is designed to investigate the efficacy and safety of S-1 alone, an oral pyrimidine fluoride, to which an indication of "inoperable or recurrent breast cancer" was added, as a first-line therapy in patients with inoperable or recurrent breast cancer by comparing it with Capecitabine alone, which is already approved of the same indication.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-diagnosed breast cancer with metastasis in multiple organs
* Performance Status (World Health Organization :WHO) 0-2
* Functions below are maintained in major organs:

  * Leukocyte count: 4,000/mm3 to 12,000/mm3
  * Neutrophil count: >2,000/mm3 or more
  * Platelet count: <100,000/mm3 or more
  * Hemoglobin: >9.5 g/dL
  * Total bilirubin: >1.5 mg/dL
  * AST(GOT): within twice a normal upper value in an institution
  * AST(GPT): within twice a normal upper value in an institution
  * BUN: < 25 mg/dL
  * Creatinine: within a normal upper value in the institution
  * 24 hours creatinine clearance: >50 mL/min (using the Cockcroft-Gault formula)
  * Women's Ccr = Body weight x (140-Age)/(72 x Serum creatinine) x 0.85
* Written informed consent will be obtained for patients for entering this study

Exclusion Criteria:

* Patients with synchronous multiple cancers
* Complicated with infection
* Fever from suspected infection
* Metastasis to the central nerve system
* A history of ischemic cardiac diseases
* Active gastrointestinal ulcer
* Severe nerve disorder
* Women who are potentially pregnant, pregnant, or breast-feeding
* Severe drug allergy
* Severe suppression of the bone marrow
* Severe renal disorder
* Being treated with other pyrimidine fluoride antineoplastic agents (including any combination therapy)
* Being treated with flucytosine
* Complicated with the infection onset which a study doctor assesses to be inappropriate for this study

Ages: 25 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2008-04; Primary Completion 2012-07 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daigo Yamamoto, MD, Principal Investigator — Department of Surgery, Kansai Medical University Hirakata Hospital
Locations (8):
- Japan (8):
  - Seiko Hospital, Neyagawa, Osaka
  - Kyushu Central Hospital, Fukuoka
  - Kansai Medical University Hirakata Hospital, Hirakata
  - Hirosaki University Hospital, Hirosaki
  - Hiroshima University Hospital, Hiroshima
  - Shinyahashiradai Hospital, Matsudo
  - The University of Tokyo Hospital, Tokyo
  - Nagumo Clinic, Tokyo

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Capecitabine Arm | S-1 Arm
Started | 73 | 69
Completed | 71 | 65
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Capecitabine Arm | S-1 Arm | Total
Number analyzed (Participants) | 71 | 65 | 136
Age, Continuous [Median (Full Range); unit: years] | 61 [35 to 86] | 62 [33 to 83] | 62 [33 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 65 | 136
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Time Frame: The follow up period will be two years after the last dose has been administered.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Capecitabine Arm | S-1 Arm
Number analyzed (Participants) | 71 | 65
years | 1.2 [0.76 to 2.04] | 1.3 [0.96 to 2.68]

2. Secondary Outcome: Adverse Events
Time Frame: The follow up period will be two years after the last dose has been administered.
Reporting Status: Not Posted

3. Secondary Outcome: Antitumor Effects
Time Frame: The follow up period will be two years after the last dose has been administered.
Reporting Status: Not Posted

4. Secondary Outcome: Time to Treatment Failure
Time Frame: The follow up period will be two years after the last dose has been administered.
Reporting Status: Not Posted

5. Secondary Outcome: Survival Rate
Time Frame: The follow up period will be two years after the last dose has been administered.
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Capecitabine Arm | S-1 Arm
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/65
Other Adverse Events (participants affected / at risk) | 44/71 | 45/65
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine Arm (N=71) | S-1 Arm (N=65)
Thrombocytopenia (Investigations) | 1 | 6
Nausea (Gastrointestinal disorders) | 10 | 17
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 18 | 7
Anaemia (Blood and lymphatic system disorders) | 7 | 8
Leukopenia (Investigations) | 6 | 10
Neutropenia (Investigations) | 7 | 5
Anorexia (Metabolism and nutrition disorders) | 10 | 12
Vomiting (Gastrointestinal disorders) | 4 | 4
Abdominal pain (Gastrointestinal disorders) | 5 | 3
Stomatitis (Gastrointestinal disorders) | 3 | 6
Diarrhea (Congenital, familial and genetic disorders) | 6 | 11
Transaminase (Investigations) | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes